CLINICAL TRIAL: NCT02095106
Title: Waterproof Casting for Pediatric Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mauricio Silva, Medical Director, Orthopaedic Institute for Children, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14-000218
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-09

CONDITIONS: Pediatric Distal Radius Fractures
Keywords: forearm fractures; pediatric fractures; distal radius

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional cast first (Other): Patients in this group will first receive a traditional fiberglass cast for two weeks, after which this cast will be removed and a waterproof cast applied.
  Interventions: Device: Waterproof Cast; Device: Traditional cast
- Waterproof cast first (Other): Patients in this group will receive a waterproof cast for 2 weeks, after which the waterproof cast will be removed and a traditional fiberglass cast will be applied for an additional two weeks.
  Interventions: Device: Waterproof Cast; Device: Traditional cast

INTERVENTIONS:
Device: Waterproof Cast
  Other Names: HM Cast
Device: Traditional cast
  Other Names: 3M Traditional fiberglass cast

SUMMARY:
Distal radius fractures are one of the most commonly seen fractures in children. Traditionally, minimally angulated or non-displaced distal radius fractures are treated with short or long-arm cast immobilization for up to 8 weeks. The traditional fiberglass casts used must be kept dry to prevent inflammation and potential infection. If a fiberglass cast gets wet, it must be removed and replaced. In general, waterproof casting has been shown to improve patient comfort and overall satisfaction.

We intend to explore the efficacy of a new, waterproof cast made of a hybrid mesh in the treatment of minimally angulated distal radius fractures in children using a randomized, controlled, cross-over study design. We will include patients between 4 and 14 years of age with minimally angulated distal radius fractures (<15 degrees of angulation on sagittal or coronal planes) presented to the Orthopaedic Institute for Children Urgent Care Facility within 7 days of injury. As determined by a power analysis, a total of 26 patients will be enrolled in the study.

Patients eligible for the study will be randomized into one of two equally sized (n=13) groups: patients in Group 1 will receive a short arm cast made of the waterproof hybrid mesh material and patients in Group 2 will receive a regular fiberglass cast. Both groups will follow-up at two weeks for clinical and radiological evaluation, after which they will be transitioned into a regular fiberglass cast (Group 1) or a hybrid mesh waterproof cast (Group 2) for an additional two weeks. This crossover will allow both groups to experience each type of cast. After four weeks of immobilization, patients in both groups will discontinue casting and be advised to avoid contact sports or strenuous activities until week 8.

Patients in both groups will follow up 8 weeks after initial treatment for clinical and radiological evaluation to evaluate range of motion, pain, and fracture alignment. Physical function will be evaluated at weeks 1, 2, and 4 using the Activities Scale for Kids - Performance, a validated, highly reliable, self-reported measure that assesses physical function in children between 5 and 15 years. Pain will be evaluated using the Faces Pain Scale, a validated, highly reliable scale commonly used in the pediatric population. Patient satisfaction will be measured at Weeks 1, 2, and 4, and the radiographs at Week 8 will be compared with initial radiographs to assess fracture displacement and angulation. Skin changes will be assessed at week 2 and week 4 by an independent observer blinded to the type of cast that has been removed and digital photographs will be obtained and analyzed using ImageJ Image Processing and Analysis Software to calculate the surface area of any described skin changes as a percentage of total skin area originally covered by the cast. Itching will be assessed at weeks 1, 2, and 4 using a visual analogue scale in which a horizontal line of 100 mm will be presented to the patient with "no itching" at the left end of the scale and "strongest itching" at the right end.

We hope to determine whether the new, waterproof cast can result in similar clinical outcomes and patient satisfaction for distal radius fractures as compared with the traditional fiberglass cast.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 4 and 14 years of age (open physis)
2. Patients seen at Orthopedic Institute for Children within 7 days of the original injury
3. Patients with a closed, buckle, or minimally displaced and angulated fracture (< 15 degrees of angulation on sagittal or coronal planes) of the distal radius, with or without associated distal ulnar fracture.

Exclusion Criteria:

1. Skeletally mature patients (closed physis), or patients younger than 4 or older than 14 years of age.
2. Patients with displaced distal radius fractures (at least 15 degrees of angulation on sagittal or coronal planes or bayoneted apposition)
3. Any association generalized condition that affects the forearm or wrist range of motion.
4. Patients with history of a previous injury or surgery to the contralateral forearm or wrist.
5. Patients who received previous treatment for a forearm fracture
6. Open fractures

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Silva, MD, Principal Investigator — UCLA, Orthopaedic Institute for Children
Locations (1):
- Orthopaedic Institute for Children, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Cast First: Patients in this group first received a traditional fiberglass cast for two weeks, after which this cast was removed and a waterproof cast applied.
  Waterproof Cast
  Traditional cast
- Waterproof Cast First: Patients in this group received a waterproof cast for 2 weeks, after which the waterproof cast was removed and a traditional fiberglass cast applied for an additional two weeks.
  Waterproof Cast
  Traditional cast
Period: First Intervention (14 Days)
Arm/Group | Traditional Cast First | Waterproof Cast First
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Traditional Cast First | Waterproof Cast First
Started | 14 | 13
Completed | 14 | 12
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Cast First | Waterproof Cast First | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 12 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (2.3) | 10.3 (1.7) | 9.4 (2.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Fracture Displacement at 8 Weeks Post Injury
Description: The radiographs at Week 8 were compared with initial radiographs to assess fracture displacement and angulation.
Time Frame: 8 weeks post injury
Measure: Count of Participants; unit: Participants
Groups:
- Traditional Cast: Patients in this group were assessed after wearing the traditional cast for 2 weeks, as their first or second intervention.
- Waterproof Cast: Patients in this group were assessed after wearing a waterproof cast for 2 weeks, as the first or second intervention type.
Arm/Group | Traditional Cast | Waterproof Cast
Number analyzed (Participants) | 26 | 27
Participants | 26 | 27

2. Secondary Outcome: Number of Participants Without Skin Irritation at the Time of Cast Removal (2 Weeks From Injury for First Intervention Type) and at Final Cast Removal (4 Weeks Post Injury for Second Intervention Type)
Description: Skin changes were assessed after removal of the cast by an independent observer blinded to the type of cast that had been removed, with digital photographs obtained and analyzed using Image J Image Processing and Analysis Software to calculate the surface area of any described skin changes as a percentage of total skin area originally covered by the cast.
Time Frame: 4 weeks post-injury
Measure: Count of Participants; unit: Participants
Groups:
- Traditional Cast: Patients in this group received a traditional fiberglass cast for two weeks as the first or second study intervention
- Waterproof Cast First: Patients in this group received a waterproof cast for 2 weeks, as the first or second study intervention.
Arm/Group | Traditional Cast | Waterproof Cast First
Number analyzed (Participants) | 26 | 27
Participants | 26 | 27

3. Other Pre Specified Outcome: Itchiness
Description: Itchiness was assessed using a visual analog scale at the Time of Cast Removal (2 Weeks From Injury for First Intervention Type) and at Final Cast Removal (4 Weeks Post Injury for Second Intervention Type). This scale consisted of a horizontal line of 100 mm presented to the patient, with the term "no itching" at the left end of the scale and the term "strong itching" appearing at the right end of the scale.
Time Frame: 4 weeks post-injury
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Traditional Cast | Waterproof Cast First
Number analyzed (Participants) | 26 | 27
units on a scale | 3.58 [0 to 10] | 3.2 [0 to 8]

4. Other Pre Specified Outcome: Physical Function
Description: Physical function was evaluated using the Activities Scale for Kids - Performance (ASKp) at the Time of Cast Removal (2 Weeks From Injury for First Intervention Type) and at Final Cast Removal (4 Weeks Post Injury for Second Intervention Type) - to ensure that the measurement represented only the time in which the participant received each type of intervention. The ASKp is a validated, highly reliable, self-reported measure that assesses physical function in children between 5 and 15 years. Scale ranges from 0 to 100 with higher scores representing more physical activity.
Time Frame: 4 weeks post-injury
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Traditional Cast: Patients in this group received a traditional fiberglass cast for two weeks, as the first or second study intervention.
- Waterproof Cast: Patients in this group received a waterproof cast for 2 weeks, as the first or second study intervention.
Arm/Group | Traditional Cast | Waterproof Cast
Number analyzed (Participants) | 26 | 27
units on a scale | 78.06 [31.9 to 99.2] | 85.74 [49.2 to 100]

5. Other Pre Specified Outcome: Pain
Description: Pain was evaluated at the Time of Cast Removal (2 Weeks From Injury for First Intervention Type) and at Final Cast Removal (4 Weeks Post Injury for Second Intervention Type) using the Faces Pain Scale, a validated, highly reliable scale commonly used in the pediatric population. The Faces Pain Scale is a numerical self-report measure of pain intensity developed for children to score the sensation of pain from 0-10. Pictures of 6 cartoon faces ranging from neutral expression of "no pain" (0) to "very much pain" (10). Participant is asked to point to the face that shows how much participant hurts at the time of assessment [right now].
Time Frame: 4 weeks post-injury
Measure: Mean (Full Range); unit: score
Arm/Group | Traditional Cast | Waterproof Cast
Number analyzed (Participants) | 26 | 27
score | 0.8 [0 to 3] | 0.6 [0 to 3]

6. Other Pre Specified Outcome: Patient Satisfaction
Description: Patient satisfaction with the treatment was measured at the Time of Cast Removal (2 Weeks From Injury for First Intervention Type) and at Final Cast Removal (4 Weeks Post Injury for Second Intervention Type) with a survey that was presented to the patient or parent, asking them to rate the satisfaction on a scale from 1 (less satisfied) to 100 (more satisfied).
Time Frame: 4 weeks post-injury
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Traditional Cast | Waterproof Cast First
Number analyzed (Participants) | 26 | 27
units on a scale | 83.9 [60.6 to 100] | 84.0 [22.5 to 100]

ADVERSE EVENTS:
Groups:
- Waterproof Cast: Patients in this group receives a waterproof cast for 2 weeks, as the first or second study intervention
Arm/Group | Traditional Cast | Waterproof Cast
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No